CLINICAL TRIAL: NCT01224964
Title: Development and Validation of a Sputum Biomarker mRNA Panel for the Diagnostic Work-up of Asthma 3
Acronym: BioSput-Air
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A lot of patients recruited in our center were already on montelukast treatment. It was not possible to recruit sufficient patients for the study.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, prof. dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Biomarker sputum airway study3
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Asthmatic Patients
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast (Active Comparator)
  Interventions: Drug: Montelukast
- long-acting beta2-mimetic (Active Comparator)
  Interventions: Drug: long acting beta2 mimetic

INTERVENTIONS:
Drug: Montelukast — Montelukast, 10 mg
  Arms: Montelukast
Drug: long acting beta2 mimetic — ICS+long acting beta2 agonist: twice daily
  Arms: long-acting beta2-mimetic

SUMMARY:
The main objectives of the study are:

1. To unravel the importance of molecular phenotyping in predicting the response to classical anti-asthma treatment (leukotriene antagonists)

The investigators have developed a non-invasive technique based on mRNA analysis of induced sputum that enables us to study airway inflammation in detail. This technique forms the basis for our current project based on the following hypotheses:

1. Different molecular asthma phenotypes exist: a Th2 phenotype and a non Th2 phenotype as reported by Woodruff and colleagues (Woodruff PG et al). Sputum mRNA cytokine levels can be used to diagnose Th2 asthma and discriminate this from non-Th2 asthma.
2. Based on our previous research and preliminary data that non-Th2 asthma can be further divided in Th17 asthma and Th1+Th2 asthma; besides these, a fourth group without Th2, Th17 or Th1 characteristics also exist.
3. These subgroups have different responses to anti-leukotrienes.

ELIGIBILITY:
Inclusion Criteria:

* uncontrolled persistent asthmatics on daily inhaled corticosteroids (GINA)

Exclusion Criteria:

* viral/fungal/bacterial infection +fever (<1 month)
* asthma exacerbation (<3 months)
* other respiratory disease (CF, ciliary dyskinesia,bronchiectasis)
* cardiac patients using beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
sputum cytokine mRNA | 8 weeks

SECONDARY OUTCOMES:
responsiveness to the medication | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MA Bullens, MD,PhD, Principal Investigator — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België; Sven F Seys, MSc, Study Director — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België
Locations (1):
- University Hospital of Leuven, Leuven, Vlaams-Brabant, Belgium